CLINICAL TRIAL: NCT04339387
Title: COVID-19 Risk Stratification
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Levine, Associate Physician, Brigham and Women's Hospital
Other Study IDs: 2020P000944
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Coronavirus; Coronavirus Sars-Associated as Cause of Disease Classified Elsewhere
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronavirus Disease 2019 positive, suitable for discharge: Patients with Coronavirus Disease 2019 who do not require supplemental oxygen, do not require intensive care unit-level care, and do not die.
- Coronavirus Disease 2019 positive, not suitable for discharge: Patients with Coronavirus Disease 2019 who do require supplemental oxygen, do require intensive care unit-level care, or do die.

SUMMARY:
The investigators seek to derive and validate a clinically useful risk score for patients with Coronavirus Disease 2019 to aide clinicians in the safe discharge of patients.

DETAILED DESCRIPTION:
The investigators a-priori plan the following analysis:

1. Derivation and Retrospective Validation.

   * Select all adult patients with a positive reverse transcription polymerase chain reaction for severe acute respiratory syndrome coronavirus 2 beginning March 1, 2020 until approximately 1000 patients are included.
   * Use 75% of this cohort to develop a simple risk-score that prognosticates a patient's suitability for discharge (no supplemental oxygen, no intensive care unit, and no death). Use multivariable logistic regression with forward selection informed by clinical judgement to choose variables a priori that emphasizes readily available data and easy calculation for use at the point of care.
   * Use 25% of this cohort to retrospectively validate the risk-score.
2. Prospective Validation.

   * Select all adult patients with a positive reverse transcription polymerase chain reaction for severe acute respiratory syndrome coronavirus 2 as soon as the derivation cohort in step 1 is assembled. Include approximately 250 patients.
   * Use this sample to prospectively validate the risk-score developed in part 1.

ELIGIBILITY:
Inclusion Criteria:

* Positive reverse transcription polymerase chain reaction for severe acute respiratory syndrome coronavirus 2
* Age 18 and older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes every adult patient noted positive for severe acute respiratory syndrome coronavirus 2 in the entire Partners HealthCare system, a consortium hospitals and health care entities located in Massachusetts that cares for over 1.5 million patients each year.
Sampling Method: Non-Probability Sample
Enrollment: 1326 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Suitable for discharge | Duration of participation in cohort, expected to be between 1 day and 20 days.
  Patient with COVID-19 who does not require supplemental oxygen, does not require intensive care unit-level care, and does not die.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Investigators may provide reasonable requests for IPD. These requests will be reviewed by the study team and institution on a case by case basis.